CLINICAL TRIAL: NCT05572385
Title: Clinical and Neurophysiological Features of Neurorehabilitation Effects in Cerebrovascular Aphasia
Brief Title: Clinic and Neurophysiology of Aphasia Treatment
Acronym: AphasRehab
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Klinik Bavaria (Other)
Responsible Party: Principal Investigator, Michael Adamaszek, Head Dept. Clinical and Cognitive Neurorehabilitation, Klinik Bavaria
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: EK-BR-157/20-1
Record Dates: First submitted 2022-10-04; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Aphasia, Acquired
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with aphasia (Active Comparator): Patients with a clinical aphasia (20 receptive, 20 expressive) with a specific logopedic treatment, with specific EEG measurement at start and end of treatment schedule.
  Interventions: Behavioral: CIAT + Conventional neurorehabilitative therapy
- Patients without aphasia (No Intervention): Patients with comparable stroke characteristics, but without clinical aphasia.

INTERVENTIONS:
Behavioral: CIAT + Conventional neurorehabilitative therapy — CIAT = Constrained induced aphasia therapy
  Other Names: Conventional neurorehabilitative therapy
  Arms: Patients with aphasia

SUMMARY:
In the planned study, clinical and electrophysiological features of aphasia recovery in stroke patients are investigated.

DETAILED DESCRIPTION:
Clinical neurorehabilitation faces a major challenge of functional recovery in aphasia, i.e. guiding the structural and temporal dynamics of reorganization within responsible neural networks. Here, according to current research, relevant neural factors affecting the treatment and thus the functional recovery of aphasia patients after stroke are of interest, highlighting structural as well as functional neuroanatomical features. Of particular interest are not only the functional localization of affected cerebral regions, but more the clinical and neurophysiological patterns which might help to factorize and predict the therapeutic outcome. In the planned study, the clinical and neurophysiological characteristics of the dynamics of language function recovery in relation to the intensity of professional speech therapy (constraint induced aphasia therapie - CIAT) will be recorded in 40 patients with aphasia resulting from a cerebrovascular event. The aim of this study is to test the value of neurophysiological aspects based on electroencephalographic (EEG) parameters such as event-related potentials (N400, P600, theta band activity) for the identification of specific neuronal markers, which in turn support predictive statements for individual therapy planning of logopedic treatment in neurorehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* patients with a cerebrovascular event

Exclusion Criteria:

* premorbid brain disorder

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
EEG correlates of language reconstitution | 3-6 months after stroke
  Identitification of EEG features (N400, P600, Theta band activity) that correlate with clinical outcome of language reconstitution.

IPD SHARING:
Plan to Share IPD: No